CLINICAL TRIAL: NCT03692507
Title: Effects of Nutritional Preconditioning on the Nutritional Status of Patients Undergoing Major General Surgeries and Subsequent Operative Outcomes
Brief Title: Effects of Nutritional Preconditioning on the Patient's Outcomes After Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Francisco (Other)
Collaborators: California State university, Fresno, Department of Food Science and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018006
Record Dates: First submitted 2018-06-05; First posted 2018-10-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Major Abdominal/GI Surgery
Keywords: HMB: β-hydroxy β-methylbutyrate; MNA: Mini Nutrition Assessment; GMS: Graz Malnutrition Screening; MUST: Malnutrition Universal Screening Tool; MST: Malnutrition Screening Tool; SGA: Subjective Global Assessment; REE: Resting Energy Expenditure; IC: Indirect calorimetry
MeSH Terms: interventions — Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HMB only (Experimental): Taking HMB supplements three times a day
  Interventions: Dietary Supplement: HMB
- Protein and HMB (Experimental): Drinking Ensure Enlive shakes
  Interventions: Dietary Supplement: Protein and HMB
- Current ERAS (High Protein) (Experimental): Drinking Ensure surgery shakes + Ensure pre-surgery
  Interventions: Dietary Supplement: ERAS

INTERVENTIONS:
Dietary Supplement: HMB — Patients in the first group (HMB only) will take 3 capsules of HMB by VitaMonk™ (1000mg/capsule) daily (morning, noon, and night) for 5 days prior to surgery.
  Arms: HMB only
Dietary Supplement: Protein and HMB — Patients in the second group (HMB + protein) will drink 2- 8oz bottles of Ensure Enlive daily (morning and night) for 5 days prior to surgery. Each bottle contains 1500mg of HMB and 20 g of protein.
  Arms: Protein and HMB
Dietary Supplement: ERAS — Patients in the third group (High protein) will drink 2- 8oz bottles of Ensure surgery daily (morning and night) for 5 days prior to surgery. Each bottle contains 18g of protein. and a clear 50g Pre-surgery drink on the day of surgery
  Other Names: Protein
  Arms: Current ERAS (High Protein)

SUMMARY:
Malnutrition is a serious problem in patients undergoing major surgeries and has a direct association with increased morbidity, mortality, length of stay (LOS), increased readmissions and cost of care. Studies suggest several advantages of supplementation with protein or specific amino acids in malnourished patients. Dietary leucine or its metabolite β-hydroxy β-methylbutyrate (HMB) can improve skeletal muscle mass and function by increasing transcriptional level of protein synthase, while other high protein or amino acids like Glutamine or Arginine supplements only provide protein-amino acids pool for patients while body's preferred fuel during metabolic stress is endogens protein, rather than exogenous diet.

In this study the investigators seek to achieve two distinct goals:

1. Determine the patients' nutritional status before and after major surgeries by baseline and subsequent nutritional assessments, according to ASPEN's criteria. In addition, the investigators were going to use indirect calorimetry to determine the Resting Energy Expenditure (REE) in different phases of pre- and postoperative periods. The investigators also propose to compare different serum protein markers and their ratios in order to correlate them with ASPEN's criteria for nutritional status quantification. In Summary, three discrete tools including ASPEN's criteria, indirect calorimetry, and serum biomarkers are going to be used in conjunction with each other to delineate the patients' nutritional status in various pre- and post-operative periods.
2. Patients undergoing major surgeries were supplemented with high protein with ß-hydroxy ß-methylbutyrate (HMB) (Ensure, Envile) or HMB only as a control, in order to improve their nutritional status and improve postoperative outcomes. The investigators looked for depict meaningful improvements in surgical outcomes by nutritional supplementation with or without HMB.

DETAILED DESCRIPTION:
Hypotheses:

We hypothesize that patients receiving high protein nutritional supplementation with HMB (Ensure Enlive) will have meaningful improvements in surgical outcomes rather than if they receive HMB only. Also, by comparing different methods of malnutrition designation, we are hypothesizing that by conduction this study, we will have a better understanding of malnutrition and its consequences in the Central Valley of California. Furthermore, we are planning to improve patient outcomes and significantly reduce the health care costs of the Valley by proper nutritional supplementation.

Specific Aims:

Demonstrate the important role β-hydroxy β-methyl butyrate (HMB) supplementation with or without high protein nutrition supplement in patients undergoing major surgeries and their outcomes.

Develop the current ERAS protocol used in Community Regional Medical Center by determining the best oral nutrition supplement prior to surgery Emphasize the importance of using oral nutrition supplements before major surgeries to decrease the patient's recovery after surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Dr. Amir Fathi as attending surgeon
* Adult patients (age >18) undergoing major abdominal and GI surgeries
* Patients at risk for malnutrition based on the ASPEN and The Academy malnutrition criteria

Exclusion Criteria:

* Pediatric patients
* Patients undergoing chemotherapy or radiation
* Patients with known allergies to products (Ensure Enlive, HMB)
* Patients that are unable to comply with all requirements
* Vegan patients
* Pregnant patients
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-30 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Patient length of hospital stay | day seven and day thirty after surgery
  Length of hospital stay (LOS) will be measured for all participating patients. Average LOS in the intervention group will be compared with the average LOS in the control group.

SECONDARY OUTCOMES:
Change in transcriptional key proteins expression level | one year
  Western blot analysis of muscle obtained at biopsy from patients

CONTACTS AND LOCATIONS:
Overall Officials: Amir h Fathi, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Community Regional Medical Center, Fresno, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Studley HO. Percentage of weight loss: a basic indicator of surgical risk in patients with chronic peptic ulcer. 1936. Nutr Hosp. 2001 Jul-Aug;16(4):141-3; discussion 140-1. No abstract available. PMID 11680474
- [Background] Fairfield KM, Askari R, Lipman TO, Sanfey H, Collins KA. Overview of perioperative nutritional support. UpToDate. Last full review/revision: September. 2014
- [Background] Mueller C, Compher C, Ellen DM; American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.) Board of Directors. A.S.P.E.N. clinical guidelines: Nutrition screening, assessment, and intervention in adults. JPEN J Parenter Enteral Nutr. 2011 Jan;35(1):16-24. doi: 10.1177/0148607110389335. No abstract available. PMID 21224430
- [Background] Corkins MR, Guenter P, DiMaria-Ghalili RA, Jensen GL, Malone A, Miller S, Patel V, Plogsted S, Resnick HE; American Society for Parenteral and Enteral Nutrition. Malnutrition diagnoses in hospitalized patients: United States, 2010. JPEN J Parenter Enteral Nutr. 2014 Feb;38(2):186-95. doi: 10.1177/0148607113512154. Epub 2013 Nov 18. PMID 24247093
- [Background] Gomes F, Emery PW, Weekes CE. Risk of Malnutrition Is an Independent Predictor of Mortality, Length of Hospital Stay, and Hospitalization Costs in Stroke Patients. J Stroke Cerebrovasc Dis. 2016 Apr;25(4):799-806. doi: 10.1016/j.jstrokecerebrovasdis.2015.12.017. Epub 2016 Jan 18. PMID 26796058
- [Background] McWhirter JP, Pennington CR. Incidence and recognition of malnutrition in hospital. BMJ. 1994 Apr 9;308(6934):945-8. doi: 10.1136/bmj.308.6934.945. PMID 8173401
- [Background] Gavazzi C, Colatruglio S, Valoriani F, Mazzaferro V, Sabbatini A, Biffi R, Mariani L, Miceli R. Impact of home enteral nutrition in malnourished patients with upper gastrointestinal cancer: A multicentre randomised clinical trial. Eur J Cancer. 2016 Sep;64:107-12. doi: 10.1016/j.ejca.2016.05.032. Epub 2016 Jul 5. PMID 27391922
- [Background] Keller H, Allard J, Vesnaver E, Laporte M, Gramlich L, Bernier P, Davidson B, Duerksen D, Jeejeebhoy K, Payette H. Barriers to food intake in acute care hospitals: a report of the Canadian Malnutrition Task Force. J Hum Nutr Diet. 2015 Dec;28(6):546-57. doi: 10.1111/jhn.12314. Epub 2015 Apr 20. PMID 25891798
- [Background] Gropper SS, Smith JL. Advanced nutrition and human metabolism: Cengage Learning; 2012.
- [Background] Schlein KM, Coulter SP. Best practices for determining resting energy expenditure in critically ill adults. Nutr Clin Pract. 2014 Feb;29(1):44-55. doi: 10.1177/0884533613515002. Epub 2013 Dec 12. PMID 24336442
- [Background] Burden S, Todd C, Hill J, Lal S. Pre-operative nutrition support in patients undergoing gastrointestinal surgery. Cochrane Database Syst Rev. 2012 Nov 14;11:CD008879. doi: 10.1002/14651858.CD008879.pub2. PMID 23152265
- [Background] McClave SA, Martindale RG, Kiraly L. The use of indirect calorimetry in the intensive care unit. Curr Opin Clin Nutr Metab Care. 2013 Mar;16(2):202-8. doi: 10.1097/MCO.0b013e32835dbc54. PMID 23340008
- [Background] Fraipont V, Preiser JC. Energy estimation and measurement in critically ill patients. JPEN J Parenter Enteral Nutr. 2013 Nov;37(6):705-13. doi: 10.1177/0148607113505868. Epub 2013 Oct 10. PMID 24113283
- [Background] Roller RE, Eglseer D, Eisenberger A, Wirnsberger GH. The Graz Malnutrition Screening (GMS): a new hospital screening tool for malnutrition. Br J Nutr. 2016 Feb 28;115(4):650-7. doi: 10.1017/S0007114515004924. Epub 2015 Dec 14. PMID 26652856
- [Background] Karsegard VL, Ferlay O, Maisonneuve N, Kyle UG, Dupertuis YM, Genton L, Pichard C. [Simplified malnutrition screening tool: Malnutrition Universal Screening Tool (MUST)]. Rev Med Suisse Romande. 2004 Oct;124(10):601-5. French. PMID 15573502
- [Background] Poulia KA, Yannakoulia M, Karageorgou D, Gamaletsou M, Panagiotakos DB, Sipsas NV, Zampelas A. Evaluation of the efficacy of six nutritional screening tools to predict malnutrition in the elderly. Clin Nutr. 2012 Jun;31(3):378-85. doi: 10.1016/j.clnu.2011.11.017. Epub 2011 Dec 17. PMID 22182948
- [Background] White JV, Guenter P, Jensen G, Malone A, Schofield M; Academy Malnutrition Work Group; A.S.P.E.N. Malnutrition Task Force; A.S.P.E.N. Board of Directors. Consensus statement: Academy of Nutrition and Dietetics and American Society for Parenteral and Enteral Nutrition: characteristics recommended for the identification and documentation of adult malnutrition (undernutrition). JPEN J Parenter Enteral Nutr. 2012 May;36(3):275-83. doi: 10.1177/0148607112440285. PMID 22535923
- [Background] Doweiko JP, Nompleggi DJ. The role of albumin in human physiology and pathophysiology, Part III: Albumin and disease states. JPEN J Parenter Enteral Nutr. 1991 Jul-Aug;15(4):476-83. doi: 10.1177/0148607191015004476. PMID 1895489
- [Background] Felder S, Braun N, Stanga Z, Kulkarni P, Faessler L, Kutz A, Steiner D, Laukemann S, Haubitz S, Huber A, Mueller B, Schuetz P. Unraveling the Link between Malnutrition and Adverse Clinical Outcomes: Association of Acute and Chronic Malnutrition Measures with Blood Biomarkers from Different Pathophysiological States. Ann Nutr Metab. 2016;68(3):164-72. doi: 10.1159/000444096. Epub 2016 Feb 9. PMID 26855046
- [Background] Marcason W. Malnutrition: where do we stand in acute care? J Acad Nutr Diet. 2012 Jan;112(1):200. doi: 10.1016/j.jand.2011.11.003. Epub 2011 Dec 22. No abstract available. PMID 22709647
- [Background] Tan CS, Read JA, Phan VH, Beale PJ, Peat JK, Clarke SJ. The relationship between nutritional status, inflammatory markers and survival in patients with advanced cancer: a prospective cohort study. Support Care Cancer. 2015 Feb;23(2):385-91. doi: 10.1007/s00520-014-2385-y. Epub 2014 Aug 13. PMID 25112562
- [Background] Tappenden KA, Quatrara B, Parkhurst ML, Malone AM, Fanjiang G, Ziegler TR. Critical role of nutrition in improving quality of care: an interdisciplinary call to action to address adult hospital malnutrition. JPEN J Parenter Enteral Nutr. 2013 Jul;37(4):482-97. doi: 10.1177/0148607113484066. Epub 2013 Jun 4. PMID 23736864
- [Background] He X, Duan Y, Yao K, Li F, Hou Y, Wu G, Yin Y. beta-Hydroxy-beta-methylbutyrate, mitochondrial biogenesis, and skeletal muscle health. Amino Acids. 2016 Mar;48(3):653-664. doi: 10.1007/s00726-015-2126-7. Epub 2015 Nov 14. PMID 26573541
- [Background] Inaba M, Terai H, Nakajima Y, et al. Usefulness of oral administration of the specialized amino acid supplement consisting of β-hydroxy-β-methylbutyrate, L-arginine and L-glutamine (Abound™) for chronic soft tissue diseases in the mouth. SDRP Journal of Food Science & Technology. 2016;1.
- [Background] Deutz NE, Pereira SL, Hays NP, Oliver JS, Edens NK, Evans CM, Wolfe RR. Effect of beta-hydroxy-beta-methylbutyrate (HMB) on lean body mass during 10 days of bed rest in older adults. Clin Nutr. 2013 Oct;32(5):704-12. doi: 10.1016/j.clnu.2013.02.011. Epub 2013 Mar 4. PMID 23514626
- [Background] Lowery RP, Joy JM, Rathmacher JA, Baier SM, Fuller JC Jr, Shelley MC 2nd, Jager R, Purpura M, Wilson SM, Wilson JM. Interaction of Beta-Hydroxy-Beta-Methylbutyrate Free Acid and Adenosine Triphosphate on Muscle Mass, Strength, and Power in Resistance Trained Individuals. J Strength Cond Res. 2016 Jul;30(7):1843-54. doi: 10.1519/JSC.0000000000000482. PMID 24714541
- [Background] Ekinci O, Yanik S, Terzioglu Bebitoglu B, Yilmaz Akyuz E, Dokuyucu A, Erdem S. Effect of Calcium beta-Hydroxy-beta-Methylbutyrate (CaHMB), Vitamin D, and Protein Supplementation on Postoperative Immobilization in Malnourished Older Adult Patients With Hip Fracture: A Randomized Controlled Study. Nutr Clin Pract. 2016 Dec;31(6):829-835. doi: 10.1177/0884533616629628. Epub 2016 Jul 9. PMID 26965178
- [Background] Wilson JM, Lowery RP, Joy JM, Walters JA, Baier SM, Fuller JC Jr, Stout JR, Norton LE, Sikorski EM, Wilson SM, Duncan NM, Zanchi NE, Rathmacher J. beta-Hydroxy-beta-methylbutyrate free acid reduces markers of exercise-induced muscle damage and improves recovery in resistance-trained men. Br J Nutr. 2013 Aug 28;110(3):538-44. doi: 10.1017/S0007114512005387. Epub 2013 Jan 3. PMID 23286834
- [Background] Bollhalder L, Pfeil AM, Tomonaga Y, Schwenkglenks M. A systematic literature review and meta-analysis of randomized clinical trials of parenteral glutamine supplementation. Clin Nutr. 2013 Apr;32(2):213-23. doi: 10.1016/j.clnu.2012.11.003. Epub 2012 Nov 9. PMID 23196117
- [Background] Heyland D, Muscedere J, Wischmeyer PE, Cook D, Jones G, Albert M, Elke G, Berger MM, Day AG; Canadian Critical Care Trials Group. A randomized trial of glutamine and antioxidants in critically ill patients. N Engl J Med. 2013 Apr 18;368(16):1489-97. doi: 10.1056/NEJMoa1212722. PMID 23594003
- [Background] Gade J, Levring T, Hillingso J, Hansen CP, Andersen JR. The Effect of Preoperative Oral Immunonutrition on Complications and Length of Hospital Stay After Elective Surgery for Pancreatic Cancer--A Randomized Controlled Trial. Nutr Cancer. 2016;68(2):225-33. doi: 10.1080/01635581.2016.1142586. Epub 2016 Mar 4. PMID 26943500
- [Background] Evans DC, Martindale RG, Kiraly LN, Jones CM. Nutrition optimization prior to surgery. Nutr Clin Pract. 2014 Feb;29(1):10-21. doi: 10.1177/0884533613517006. Epub 2013 Dec 17. PMID 24347529
- [Background] Bozkirli BO, Gundogdu RH, Ersoy E, Lortlar N, Yildirim Z, Temel H, Oduncu M, Karakaya J. Pilot Experimental Study on the Effect of Arginine, Glutamine, and beta-Hydroxy beta-Methylbutyrate on Secondary Wound Healing. JPEN J Parenter Enteral Nutr. 2015 Jul;39(5):591-7. doi: 10.1177/0148607113520433. Epub 2014 Jan 24. PMID 24463351
- [Background] Sun S, Reynolds J, Erceg DN, et al. Validation Of The ReeVue (TM) And CardioCoachCo2 (TM) Metabolic Systems For Measuring Resting Energy Expenditure: 1525: Board# 127 May 27 9: 30. 2009.